CLINICAL TRIAL: NCT04386577
Title: Effects of Vitamin D and Omega-3 Supplementation on Telomeres in VITAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Augusta University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Yanbin Dong, Regents Professor, Augusta University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016p001917; R01HL131674-01 (NIH)
Record Dates: First submitted 2017-08-15; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Aging
Keywords: vitamin D, omega-3 fatty acid, telomere length, inflammation
MeSH Terms: conditions — Inflammation | interventions — Cholecalciferol; Fish Oils; Fatty Acids, Omega-3

STUDY DESIGN:
Intervention Model Description: VITAL is a 2 x 2 factorial randomized, double-blind, placebo-controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D + fish oil (Active Comparator): Dietary supplement: Vitamin D3 (cholecalciferol), 2000 IU per day. Drug: Omega-3 fatty acids (fish oil), Omacor, 1 capsule per day. Each capsule contains 840 mg of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid (EPA) and 375 mg of docosahexaenoic acid (DHA).
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol); Drug: fish oil
- Vitamin D + fish oil placebo (Active Comparator): Dietary supplement: Vitamin D3 (cholecalciferol), 2000 IU per day. Dietary supplement: Fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)
- Vitamin D placebo + fish oil (Active Comparator): Drug: Omega-3 fatty acids (fish oil), Omacor, 1 capsule per day. Dietary supplement: Vitamin D3 placebo
  Interventions: Drug: fish oil
- Vitamin D placebo + fish oil placebo (Placebo Comparator): Dietary supplement: Vitamin D3 placebo Dietary supplement: Fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol); Drug: fish oil

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol) — Eligible participants were assigned by chance to one of four groups: (1) daily vitamin D3 and omega-3; (2) daily vitamin D3 and omega-3 placebo; (3) daily vitamin D placebo and omega-3; or (4) daily vitamin D placebo and omega-3 placebo. At baseline, year 2 and year 4 of the trial, a subcohort of 1,054 VITAL participants living within driving distance of Boston, Massachusetts received detailed in-clinic health assessments at the Clinical and Translational Science Center (CTSC) of Brigham and Women's Hospital. During CTSC visits, participants have a clinical exam, including measurement of height, weight, other anthropometrics, blood pressure, and physical performance. They also provide fasting blood and urine samples, and undergo 2-hour oral glucose tolerance testing, lung function testing (spirometry), electrocardiograms, bone mineral density testing, 2D-echocardiography, and assessments of thinking and mood.
  Arms: Vitamin D + fish oil; Vitamin D + fish oil placebo; Vitamin D placebo + fish oil placebo
Drug: fish oil — Eligible participants were assigned by chance to one of four groups: (1) daily vitamin D3 and omega-3; (2) daily vitamin D3 and omega-3 placebo; (3) daily vitamin D placebo and omega-3; or (4) daily vitamin D placebo and omega-3 placebo. At baseline, year 2 and year 4 of the trial, a subcohort of 1,054 VITAL participants living within driving distance of Boston, Massachusetts received detailed in-clinic health assessments at the Clinical and Translational Science Center (CTSC) of Brigham and Women's Hospital. During CTSC visits, participants have a clinical exam, including measurement of height, weight, other anthropometrics, blood pressure, and physical performance. They also provide fasting blood and urine samples, and undergo 2-hour oral glucose tolerance testing, lung function testing (spirometry), electrocardiograms, bone mineral density testing, 2D-echocardiography, and assessments of thinking and mood.
  Other Names: Omega-3 fatty acid
  Arms: Vitamin D + fish oil; Vitamin D placebo + fish oil; Vitamin D placebo + fish oil placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) was a randomized clinical trial in 25,871 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or fish oil (1 gram of omega-3 fatty acids) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study is being conducted among participants in VITAL-CTSC cohort and will examine whether vitamin D or fish oil supplementation has beneficial effects on cellular aging.

DETAILED DESCRIPTION:
This project is an ancillary study based on the parental study "the VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259)" at the Harvard Clinical and Translational Science Centre (CTSC) and Brigham and Women's Hospital. Our research focuses on the separate and synergistic effects of vitamin D and omega -3 supplements on telomere length, a cellular aging marker, using de-identified samples from VITAL-CTSC cohort.

Aims: 1) To test the hypothesis that vitamin D supplementation decreases leukocyte telomere length attrition. The investigators will determine the effect of vitamin D supplementation on telomere length attrition over time (Baseline, Year 2, and Year 4); 2) To test the hypothesis that marine omega-3 fatty acid supplementation decreases LTL attrition. The investigators will determine the effect of marine omega-3 fatty acid supplementation on telomere length attrition over time (Baseline, Year 2, and Year 4); 3) To determine to what extent the effects of vitamin D or omega-3 supplementation on inflammatory cytokines and CVD risk factors are mediated by telomere length attrition over time; 4) To explore the synergistic effects vitamin D and omega-3 fatty acid supplementation.

ELIGIBILITY:
Inclusion Criteria:

The subcohort of 1,054 participants in VITAL (NCT 01169259) who are receiving detailed health assessments at a Clinical and Translation Science Center at Boston are eligible to participate in this ancillary study:

-

Exclusion Criteria: None

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1054 (Actual)
Dates: Start 2016-08-19 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in telomere length | 4 years
  Leukocyte telomere length (LTL) will be measured using quantitative polymerase chain reaction method at the baseline, year 2 and year 4. we will examine the effect of randomization to vitamin D (primary Aim 1 and or fish oil (primary Aim 2) compared o placebo is different over time on changes in telomere length.

SECONDARY OUTCOMES:
Changes in Inflammation markers | 4 years
  We will examine the changes in plasma markers of inflammation (CRP, interleukin-6 (IL-6), interleukin-10 (IL-10), interleukin-12 (IL-12), tumor necrosis factor-alpha (TNF-a) in plasma samples collected at the baseline, year 2 and year 4. We will
  examine whether change in LTL is a mediator of change of inflammatory and cardiovascular disease (CVD) risk.

CONTACTS AND LOCATIONS:
Overall Officials: Yanbin Dong, MD, PhD, Principal Investigator — Augusta University
Locations (1):
- Georgia Prevention Institute, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators recognize and fully support the principles of resource and data sharing that have been endorsed by the NIH. Since VITAL is a randomized, double-blind, placebo-controlled trial, the investigators will not be able to share any unblinded data involving randomized treatments with internal or outside investigators while the trial in ongoing (with the exception of the Independent Data and Safety Monitoring Board). However, the investigators will maintain our strong commitment to the full communication of important study results to participants and the scientific community through rapid publication of primary findings, presentations at major meetings, as well as through appropriate lay interviews and lay publications.